CLINICAL TRIAL: NCT06523647
Title: Clinical Efficacy of Ustekinumab in Crohn's Disease: an Observational Study With Retrospective and Prospective Components
Brief Title: Clinical Efficacy of Ustekinumab in Crohn's Disease
Status: Recruiting | Type: Observational
Sponsor: Kazakhstan Scientific Society for Study of intestine diseases (Other)
Responsible Party: Sponsor
Other Study IDs: KSSSID-01-23
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Clinical Efficacy of Ustekinumab in Crohn's Disease: an Observational Study With Retrospective and Prospective Components.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older;
* Patients who were first prescribed Ustekinumab between January 1 and December 31, 2024
* Patients who provided written informed consent to participate in the study

Exclusion Criteria:

* Contraindications to the use of the drug Ustekinumab per the current instructions:

  * Clinically significant active infection (active tuberculosis, active viral hepatitis);
  * Pregnancy and lactation;
  * A history of clinically significant, in the opinion of the investigator, psychiatric disorders that may interfere with the study procedures and compliance with the drug regimen;
  * Ulcerative colitis;
  * Malignant gastrointestinal diseases in history or at the time of inclusion in the study;
  * Decompensated chronic diseases of the liver, kidneys, cardiovascular system, systemic vasculitis, diabetes mellitus;
  * Abuse of alcohol or psychoactive drugs within 1 year before the start of this study (as reported by the patient);
* Participation in an interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include male and female patients aged 18 years and older, with a confirmed diagnosis of Crohn's disease, on therapy with the drug Ustekinumab
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a reduced level of disease activity by 30% or more according to the Crohn's Disease Activity Index | at week 24 of therapy

SECONDARY OUTCOMES:
Proportion of patients with a 30% or more reduction in disease activity according to the Crohn's Disease Activity Index | at 12 and 52 weeks of therapy
Proportion of patients in endoscopic remission based on Simple Endoscopic Score for Crohn's Disease | at 24 and 52 weeks
Dynamics of fecal calprotectin levels | at 24 and 52 weeks
Proportion of patients with normalization of Magnetic resonance enterography based on the Magnetic Resonance Index of Activity | at 12 and 52 weeks
Dynamics of quality of life assessment based on the Short Inflammatory Bowel Disease Questionnaire | at 12, 24 and 52 weeks
Dynamics of antibody synthesis to the drug Ustekinumab | at 0/1, 24 and 52 weeks
List of medications indicated in the general scheme with Odeston | through study completion, an average of 1 year
Dynamics of assessing patient adherence to treatment using the Morisky-Green scale | at 0/1, 12, 24 and 52 weeks
Collection of information on adverse reactions and/or registration of pregnancy cases | through study completion, an average of 1 year
Dynamics of red blood cell parameters | at 24 and 52 weeks
Dynamics of hemoglobin parameters | at 24 and 52 weeks
Dynamics of platelet parameters | at 24 and 52 weeks
Dynamics of leukocyte parameters with leukocyte formula | at 24 and 52 weeks
Dynamics of erythrocyte sedimentation rate parameters | at 24 and 52 weeks
Dynamics of potassium parameters | at 24 and 52 weeks
Dynamics of sodium parameters | at 24 and 52 weeks
Dynamics of C-reactive protein parameters | at 24 and 52 weeks
Dynamics of albumin parameters | at 24 and 52 weeks
Dynamics of total protein parameters | at 24 and 52 weeks
Dynamics of serum iron parameters | at 24 and 52 weeks
Dynamics of serum iron-binding capacity parameters | at 24 and 52 weeks
Dynamics of vitamin B9 parameters | at 24 and 52 weeks
Dynamics of Nutritional Risk Index indicators | at 24 and 52 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Kazakhstan (4):
  - NJSC "West Kazakhstan Marat Ospanov Medical University", Aktobe
  - Non-Profit Joint Stock Company "Kazakh National Medical University named after S.D. Asfendiyarov", Almaty
  - State-owned public enterprise with the right of economic management "Multidisciplinary City Hospital No. 1" of the Akimat of Astana, Astana
  - State-owned public enterprise with the right of economic management "Regional Clinical Hospital" of the Health Department of the Turkestan Region, Shymkent